CLINICAL TRIAL: NCT00011804
Title: Topiramate in the Treatment of Sciatica
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 010105; 01-D-0105
Record Dates: First submitted 2001-02-28; First posted 2001-03-01 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-02

CONDITIONS: Sciatica
Keywords: Low Back Pain; Lumbar Radiculopathy; Anticonvulsants; Neuropathic Pain; Analgesia; Sciatica
MeSH Terms: conditions — Sciatica; Low Back Pain; Radiculopathy; Neuralgia; Agnosia | interventions — Topiramate

INTERVENTIONS:
Drug: Topiramate

SUMMARY:
This study will test the effectiveness of topiramate to treat pain caused by lumbar radiculopathy, or sciatica. Sciatica results from damage to the lumbar nerve roots, typically causing back pain and sharp, shooting pain down one or both legs. Although sciatica is common, there are no good treatments for it. Topiramate belongs to a group of medications commonly used to treat pain caused by nerve damage.

Patients between 18 and 75 years of age who have had sciatica pain daily for at least 3 months may be eligible for this study. (This is taken from the first paragraph of the Qualification Criteria in the consent form. The inclusion criteria on page 6 of the protocol say "low back pain of 3 months duration or longer present at least 5 out of 7 days a week" and signs and symptoms of lumbar radiculopathy. Which is correct?)

Participants will provide a medical history, as well as occupational and social information. They will undergo a standard neurological examination, including a test of cognitive (thinking) abilities, muscular function, reflexes and a sensory examination. The latter involves testing with a pin placed on the surface of the skin. Participants will also have routine blood tests and will fill out questionnaires on their daily functioning and psychological well being. Additional procedures may include magnetic resonance imaging (MRI) scans and possible referral to a psychiatrist for evaluation of depression or emotional difficulties.

This "cross-over" study consists of two parts. In one part, patients will receive topiramate and in the other, an active placebo. An active placebo is a drug that does not work for the problem being studied but whose side effects are like those of the test drug. Diphenhydramine (Benadryl) is the active placebo used in this study. Diphenhydramine is an allergy medication with very mild side effects, such as drowsiness. During both parts of the study-topiramate and placebo-patients will keep a daily log in which they rate their pain, record other procedures they undergo, such as injections and manipulations, and record medication side effects.

In the first week of the study, patients will remain on their current medications and record pain levels once a day. After the first week, they will begin taking the study drugs-either topiramate in increasing doses ranging from 50 to 400 mg. or diphenhydramine in doses ranging from 6.25 to 50 mg. The drug doses will be increased gradually over 4 weeks to minimize possible side effects. Increases will continue until the maximum tolerated dose is reached. Patients will continue on the highest tolerated dose for two weeks and then be tapered off gradually over 12 days. They will remain off drugs completely for a 2-day washout period and then begin the next treatment. Those who took topiramate for the first part will take diphenhydramine for the second part and vice versa.

A study nurse will call patients twice a week throughout the study to check for problems and answer questions. A physician will see patients 6 weeks after the start of each treatment. During the last visit, at the end of the study, patients will repeat the questionnaires they filled out at the beginning of the study. Patients and their doctors will be informed of the medications that were effective in each individual's care.

DETAILED DESCRIPTION:
Irritation or damage to lumbar nerve roots referred to as lumbar radiculopathy or sciatica is a very common clinical entity with a lifetime prevalence of 1-3% in the adult population. Lumbar radiculopathy typically causes back pain and sharp, shooting pain in the leg(s). Despite its prevalence and disabling characteristics, sciatica has never been selectively studied in drug trials. We propose to study the anti-epileptic drug topiramate, which combines multiple potential analgesic actions including sodium channel blockade, GABA agonist-like effects and AMPA/kainate glutamate receptor blockade. Patients will include men and women of all ethnic backgrounds between the ages of 18 and 75 who have had signs and symptoms of sciatica for 3 months or more.

The design is a double-blind, two period cross-over study comparing topiramate to placebo. Patients will be called twice a week to individually titrate doses of topiramate towards a maximum of 800 mg per day and monitor side effects. The primary outcome measures in this study will be the daily pain scores in the low back, in the leg and combined. Patients' quality of life and activities of daily living will be secondary outcome measures as assessed by the SF 36, Oswestry, and Beck questionnaires. Sixty five patients will be enrolled in this study and the duration of the study will be 17 weeks, including one week baseline, four week escalation, two week maintenance and two week wash out for topiramate and placebo respectively.

ELIGIBILITY:
INCLUSION CRITERIA:

Low back pain of 3 months duration or longer present at least 5 out of 7 days a week are eligible.

Age between18-75 at the start of the study.

Men and women of all ethnicities.

Signs and symptoms of lumbar radiculopathy.

Ability to understand the study measures and mentally capable of giving consent to participate in the study.

Willingness to refrain from making changes in non-study medications taken for sciatica.

Patients with failed back syndrome who satisfy the following criteria:

Presence of low back pain and pain in one or both lower extremities (buttock and below) for 3 months or greater and at least one of the following:

1. Sharp and shooting pain below the knee in one or both legs.
2. Electromyographic evidence of 4th or 5th lumbar roots (L4 or L5) / first sacral root (S1) irritation on the affected side.
3. Imaging (MRI or CT/Myelogram) evidence of nerve root compression in lower lumbar region on the affected side.
4. Evidence of decreased/absent ankle reflex on the affected side.
5. Evidence of weakness of muscles below the knee on the affected side.
6. Evidence of sensory loss in L5/S1 distribution on the affected side.

Pain level of at least 4/10 on average on a scale of 0 to 10 for the past month.

EXCLUSION CRITERIA:

Hepatic and renal dysfunction (liver function tests: ALT/AST greater than 1.2 times upper limit of normal; Creatinine greater than 1.5 times upper limits of normal).

Pregnancy or lactation.

History of seizures.

Presence of pain of greater intensity in any other location than the low back or the leg.

History of narcotic abuse and/or drug or alcohol abuse in the past year.

History of fibromyalgia.

History of spinal unstability.

Cognitive impairment such that the individual is unable to give informed consent, complete study data collection tools or required study visits.

Unwillingness to use adequate contraception excluding oral contraceptive medications (such as barrier methods with spermacide simultaneously) for women.

Presence of other medical condition presenting with numbness and pain in lower extremities, such as diabetic polyneuropathy and peripheral vascular disease.

Allergy to topiramate.

Participants must not use digoxin, probenicid, carbonic anhydrase inhibitors given their possible drug interaction with topiramate.

History of nephrolithiasis.

Allergy to diphenhydramine.

History of narrow angle glaucoma.

History of asthma and COPD.

Urinary retention of any etiology.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65
Dates: Start 2001-02; Study Completion 2005-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Watson CP. The treatment of neuropathic pain: antidepressants and opioids. Clin J Pain. 2000 Jun;16(2 Suppl):S49-55. doi: 10.1097/00002508-200006001-00009. PMID 10870740
- [Background] Coderre TJ, Katz J, Vaccarino AL, Melzack R. Contribution of central neuroplasticity to pathological pain: review of clinical and experimental evidence. Pain. 1993 Mar;52(3):259-285. doi: 10.1016/0304-3959(93)90161-H. PMID 7681556
- [Background] Bajwa ZH, Sami N, Warfield CA, Wootton J. Topiramate relieves refractory intercostal neuralgia. Neurology. 1999 Jun 10;52(9):1917. doi: 10.1212/wnl.52.9.1917. No abstract available. PMID 10371550